CLINICAL TRIAL: NCT05267639
Title: Clinical Outcomes With Passive MPKs vs. Powered Prosthetic Knees by K4-level Transfemoral Amputees
Brief Title: Clinical Outcomes With Passive MPKs vs. Powered Prosthetic Knees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liberating Technologies, Inc. (Industry)
Collaborators: Hanger Clinic: Prosthetics & Orthotics (Other)
Responsible Party: Principal Investigator, Jennifer Johansson, Principal Investigator, Liberating Technologies, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20216190
Record Dates: First submitted 2021-12-09; First posted 2022-03-04 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Amputation; Amputation; Traumatic, Leg, Lower; Limb; Absence, Congenital, Lower; Prosthesis User; Lower Limb Amputation Above Knee (Injury); Amputation; Traumatic, Leg: Thigh, Between Hip and Knee
Keywords: amputee; lower limb amputee; transfemoral amputee; prosthetic knee; power knee; microprocessor knee; MPK; Ossur; lower limb prosthesis user
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants will take home two interventional devices for data collection and feedback. One of the interventions will be their usual microprocessor knee to collect as a control, and the other will be the commercially available Ossur Power Knee. Participants will be trained on the interventional knees during the first month of at-home use. Functional outcome measures and self-report surveys will also be completed in-lab before and after each take-home intervention, as well as at the last training visit, in order to form a detailed comparison between the two interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (MPK) (No Intervention): The subject will wear their usual Microprocessor Knee (MPK) for 3 months, as well as in the lab to complete outcome measures.
- Power Knee (Experimental): The subject will wear the Ossur PK in place of their usual MPK for 3 months, as well as in the lab to complete outcome measures.
  Interventions: Device: Power Knee

INTERVENTIONS:
Device: Power Knee — Newest version of the commercially-available Power Knee developed by Ossur.
  Other Names: Ossur Power Knee; Ossur Power Knee III; PK; PK3
  Arms: Power Knee

SUMMARY:
The goal of this proposed project is to gather community-based data from the K4-level Transfemoral Amputee (TFA) population to aid in evidence-based prescription of powered prosthetic knees (i.e., choosing the right device to maximize the benefit for each patient). The investigators envision that this Level 1 submission will transition into a larger follow-on Level 2 trial that will explore a larger spectrum of patient populations (K2-K4), as well as testing additional Power Knees currently in development that are expected to become commercialized in the near future. The investigators intend to use this Level 2 trial data to guide the implementation of effective prescriptions towards those that can benefit most from a given device and limit prescription to those who would not see benefit in order to ensure the most judicious use of Department of Defense (DoD) and Veteran's Affairs healthcare dollars. The findings will also be shared with the research community to help drive the design of future devices by identifying what features and functions are most beneficial to which patient populations when the devices are used outside of the laboratory. In summary, more community-based data on how powered prosthetic knees compare with MPKs is needed to allow for improved clinical decision making and clinical outcomes.

DETAILED DESCRIPTION:
The goal of this proposed project is to gather community-based data from the K4-level Transfemoral Amputee (TFA) population to aid in evidence-based prescription of powered prosthetic knees (i.e., choosing the right device to maximize the benefit for each patient). The investigators envision that this Level 1 submission will transition into a larger follow-on Level 2 trial that will explore a larger spectrum of patient populations (K2-K4), as well as testing additional Power Knees currently in development that are expected to become commercialized in the near future. The investigators intend to use this Level 2 trial data to guide the implementation of effective prescriptions towards those that can benefit most from a given device and limit prescription to those who would not see benefit in order to ensure the most judicious use of Department of Defense (DoD) and Veteran's Affairs healthcare dollars. The findings will also be shared with the research community to help drive the design of future devices by identifying what features and functions are most beneficial to which patient populations when the devices are used outside of the laboratory. In summary, more community-based data on how powered prosthetic knees compare with MPKs is needed to allow for improved clinical decision making and clinical outcomes.

This study will focus on investigating the tradeoffs between the commercially available Ossur Power Knee and traditional MPKs to identify the prosthetic knee that is best suited for K4 users during different tasks. The investigators will assess measured, observed, and self-reported outcomes achieved through real-world use of the prosthetic knees.

The results of this study will (1) provide initial data to inform the evidence-based prescription and use of powered knee technologies for K4-level individuals with sound scientific data, (2) provide pilot data for a larger clinical trial to further inform the evidence-based prescription of powered knee technologies to other K-levels to maximize patient benefit while optimizing device cost and thereby influencing clinical practice and informing policy decisions, and (3) provide data that can be disseminated to other researchers to inform the design of future powered prosthetic knees by understanding the needs of users and identifying the features and functions that are most valuable to this patient population as well as the capabilities and limitations of current devices.

The primary outcome measures for each aim are outlined as follows:

* [Mobility Primary Outcome]: daily number of steps taken
* [Safety Primary Outcome]: Activities-Specific Balance Scale
* [Wellbeing Primary Outcome]: PEQ-Well-Being (PEQ-WB)

The exploratory data collected in the in-clinic and take-home portions of this study will include number of steps and number of self-reported falls, and a series of standard outcomes measures, such as: 6MWT, SAI, RAI, PROMIS-PF short form, PLUS-M, TUG, ABC, RPE, PROMIS-Fat, fall count, PROMIS-29, ODI, PEQ-WB, and PROMIS-APSRA short form.

The investigators plan to perform a pilot longitudinal randomized crossover study to compare the powered knee and passive microprocessor knees in individuals with unilateral transfemoral amputation. The two interventions, or conditions, to be tested are: (A) Ossur PK and (B) a standard MPK. For this study the investigators will recruit individuals who are currently MPK users; therefore, for the MPK condition, they will wear their usual prosthesis (e.g. Otto Bock C-leg, Össur Rheo, etc) as they represent the current standard of care. This will be recorded as a potential confounder in post-hoc analysis. Each participant will be provided with prosthetic knees for the powered knee condition.

The order these conditions are tested in will be randomized across subjects. Block randomization using a previously developed custom software based on random number generation will be used to equally distribute the subjects into the 2 possible intervention orders (AB or BA). For each condition, the subject will be trained on and acclimated to the device during the first month of the take-home period, and then will continue to wear it at home after training for a total of three months per condition. There may be seasonal effects due to the timing of when the various test conditions are administered, however, the investigators plan to offset these effects with condition randomization, multiple site testing, and staggered start times.

Testing will consist of test sessions, training sessions, at-home wear of the device, and functional and self-report assessment at the end of each intervention condition. If the subject's current foot is not compatible with the Power Knee, they will be provided with a commercially available prosthetic foot for the study. In this case, the subject will be given an initial acclimation period of 1 month on the new foot before starting interventional testing.

After receiving IRB and HRPO (US Army Human Research Protection Office) approval, subjects will be recruited and screened for eligibility. If they are eligible and decide to participate, they will be scheduled for their first site visit. They will either be consented over the phone before their first site visit or at the first site visit. If over the phone, study staff will use the telephone script to confirm eligibility and guide the subject through consent form details. Subjects will be provided the informed consent form to read through entirely before signing, and are encouraged to ask questions at any time.

Prior to each condition, each subject will be fit and aligned on the knee by a trained certified prosthetist. An activity monitor (such as the GeneActiv™) will be worn by the subject. As the investigators have done in prior studies, the investigators will use the activity monitor to track the number of steps the subjects take in each condition. Each subject will wear the same foot for all study periods for comparability between the two knee conditions.

The subject will wear the knee being tested at home for three months. During the first month of each condition, subjects will be given time to acclimate to the knee being tested. Before and after each condition, the subject will complete a battery of outcomes and self-report surveys. Subjects will participate in at least two, but up to eight, 1 hour training sessions per knee. At a minimum, each subject will receive one training session to learn how to properly use each device for a variety of daily activities and a second session to demonstrate retention of the learned skills. The subject will continue training until they show retention of the understanding and/or proficiency of the device functions or until they have received eight training sessions, whichever comes first. After 8 training sessions, they will have completed all of the available training and will therefore continue with the study at their current proficiency level. For the powered knee condition, the investigators will work with trained and experienced clinicians, consulting prosthetic knee manufacturers as needed, to develop the training protocol and determine proficiency. At the last training session, the subject will complete a subset of the outcomes and self-report measures in order to collect and compare data from before and after the subject gets trained on each knee condition.

After the training visits are completed, subjects will be asked to continue to wear the knee full time for the remainder of the three month take-home period. Through Hanger's current patient care system, the investigators will have the ability to push out a digital to the patient's phone asking them whether they have experienced a recent fall. If they respond positively that they had a fall, follow up questions can be asked to get more specific details about the fall. After three months of at-home wear, the subject will return for the second test visit. During that visit, functional tests and self-report surveys will be administered. At the completion of the second test visit (Period 1), the subject will then be fit and aligned on the prosthetic knee condition for Period 2. The training, at home wear, and in-clinic assessments will be repeated for the next knee condition.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years old
* Unilateral transfemoral prosthesis user (limb absence between the knee and hip)
* Current user of a microprocessor-controlled knee (MPK)
* Have adequate clearance between distal end and ground for necessary knee and foot components
* Medicare Functional Classification Level (K-Level): 4
* Socket-Comfort Score: 6 or above to ensure adequate socket fit
* PLUS-M T-score of 55 or above
* Six months or more experience on a prosthesis
* Body weight between 50kg and 116kg (110lbs - 256lbs)

Exclusion Criteria:

* Present injuries to residual limb or contralateral leg affecting functional ability
* Socket issues/changes in the last 6 weeks
* Users with bone-anchored implants

Subjects can be excluded at the discretion of the investigator for other unforeseen disqualifying criteria (such as specific cognitive issues, etc.). Subjects in this study will not be discriminated by sex/gender or race/ethnicity.

Using a knee that the subject is unfamiliar with may increase the risk of falling. Therefore, pregnant women should not participate in the study and will be screened by self-disclosure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Johansson, MS, Principal Investigator — Liberating Technologies, Inc.
Locations (2):
- United States (2):
  - Liberating Technologies, Inc., Holliston, Massachusetts
  - Hanger Clinic, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Control (MPK), Then Power Knee: The subject uses their usual Microprocessor Knee (MPK) for 3 months, and then uses the Ossur Power Knee for the following 3 months.
  Power Knee: Newest version of the commercially-available Power Knee developed by Ossur.
- Power Knee, Then Control (MPK): The subject uses the Ossur PK in place of their usual MPK for 3 months, and then uses their usual Microprocessor Knee (MPK) for the following 3 months.
  Power Knee: Newest version of the commercially-available Power Knee developed by Ossur.
Period: Overall Study
Arm/Group | Control (MPK), Then Power Knee | Power Knee, Then Control (MPK)
Started | 7 | 6
Completed | 6 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (MPK), Then Power Knee | Power Knee, Then Control (MPK) | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Daily Step Count
Description: Prior to each condition, each subject will be fit and aligned on the designated knee by a trained certified prosthetist. An activity monitor (such as the GeneActiv™) will be worn by the subject for each intervention period during the final month of the condition. Similar to prior studies, the investigators will use the activity monitor to track the number of steps the subjects take in each condition per day.
  The number of steps per day are averaged over the final month in each condition. A higher value indicates a better outcome.
Time Frame: 1 Month
Population: 13 total participants. 1 participant withdrew (no data in either condition). Comparator Baseline: no data from withdrawn participant. Power Knee: step count successfully collected from 2 participants. 8 participants transitioned early and did not make it to the final month for collection. 1 activity monitor was lost in the mail. 1 file was unable to be processed/corrupt.
Measure: Mean (Standard Deviation); unit: Steps/day
Arm/Group | Control (MPK) | Power Knee
Number analyzed (Participants) | 12 | 2
Steps/day | 5747 (3212) | 3162 (1031)

2. Primary Outcome: Activities-Specific Balance Confidence Scale (ABC) - Measuring Change From Baseline
Description: Activities-specific balance confidence (ABC) scale is a structured questionnaire that measures an individual's confidence during ambulatory activities without falling or experiencing a sense of unsteadiness. It consists of 16 questions gauging the individual's confidence while doing activities, from 0 (no confidence) to 4 (complete confidence). Therefore, the total score ranges from 0 to 64, with a higher value indicating a better outcome.
  This survey will be given at the end of each study condition (2 conditions, 3 months per condition). This survey will be administered as a part of the master questionnaire.
  Analysis is reported in % of balance confidence, which is found by taking their average of all questions (sum up all questions and divide by total number of questions) and dividing that average by 4.
Time Frame: At the end of each 3 month condition
Population: 13 total enrolled. 1 participant withdrew (no data in either condition). Comparator Baseline: 1 participant withdrew from PK condition before collecting ABC. 11 analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of balance confidence
Arm/Group | Control (MPK) | Power Knee
Number analyzed (Participants) | 11 | 12
Percentage of balance confidence | 83 (17) | 83 (15)

3. Primary Outcome: PEQ-Well Being (PEQ-WB) - Measuring Change From Baseline
Description: The version of the PEQ which will be administered consists of 2 questions in 1 category (well being). For purposes of easier administration, the investigators have adopted the modified 10-point ordinal scale version of the PEQ-WB (scale 1-10, where 1 is the worst and 10 is the best relative to the questions being asked).
  This survey will be given at the end of each study condition (2 conditions, 3 months per condition). This survey will be administered as a part of the master questionnaire.
  The reported result is the average of the 2 questions in the PEQ-WB. The range of this reported result is 1-10, where a higher value indicates a better outcome.
Time Frame: At the end of each 3 month condition
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control (MPK) | Power Knee
Number analyzed (Participants) | 12 | 11
score on a scale | 8.3 (1.6) | 8.0 (1.5)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/collected during each condition. With each condition lasting about 3 months, each participant was monitored for adverse events for about 6 months total. Adverse events were monitored/assessed at least every 2 weeks by phone call, with study staff checking in more frequently if participants reached out with questions. Participants were told to reach out to study staff immediately if adverse events did occur.
Arm/Group | Control (MPK) | Power Knee
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 2/13 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (MPK) (N=13) | Power Knee (N=13)
Phantom Limb Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Participant 0102 experienced phantom limb pain and had to massage prosthetic foot with mirror therapy to help with the pain.
Broken finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Participant broke ring finger playing football and had to get an x-ray and splint.
Fall (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Participant fell while dismounting motorcycle and had bruising as well as damage to prosthesis.
Ankle swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Participant reported ankle swelling and discomfort. They received new shoes and shoe insert to address these issues

LIMITATIONS AND CAVEATS:
Limited data for the powered knee condition reduces the generalizability of these results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-08-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT05267639/Prot_002.pdf